CLINICAL TRIAL: NCT02326311
Title: Phase-III Randomized Study to Optimize TKIs Multiple Approaches - (OPTkIMA) - and Quality of Life (QoL) in Elderly Patients (≥60 Years) With Ph+ Chronic Myeloid Leukemia (CML) and MR3.0 / MR4.0 Stable Molecular Response
Brief Title: Optimization of TKIs Treatment and Quality of Life in Ph+ CML Patients ≥60 Years in Deep Molecular Response
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Prof Domenico Russo, Full Professor of Hematology, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOBSTMO-OPTKIMA-2014
Record Dates: First submitted 2014-12-17; First posted 2014-12-29 (Estimated); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Leukemia, Chronic Myeloid
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate; nilotinib; Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fixed INTERIM TKI (Active Comparator): Intervention: "fixed" intermittent administration (one month ON/one month OFF) of TKIs (imatinib, nilotinib, dasatinib)
  Interventions: Drug: imatinib; Drug: nilotinib; Drug: dasatinib
- Progressive INTERIM TKI (Experimental): Intervention: "progressive" intermittent administration (one month ON/one month OFF for the 1st year; one month ON/two months OFF for the 2nd year; one month ON/three months OFF for the 3rd year) (imatinib, nilotinib, dasatinib)
  Interventions: Drug: imatinib; Drug: nilotinib; Drug: dasatinib

INTERVENTIONS:
Drug: imatinib — Tyrosin kinase inhibitor
  Other Names: Glivec
Drug: nilotinib — Tyrosin kinase inhibitor
  Other Names: Tasigna
Drug: dasatinib — Tyrosin kinase inhibitor
  Other Names: Sprycell

SUMMARY:
In this phase III clinical randomized study, "fixed" intermittent administration (one month ON/one month OFF) of TKIs (control arm), will be compared with "progressive" intermittent administration (one month ON/one month OFF for the 1st year; one month ON/two months OFF for the 2nd year; one month ON/three months OFF for the 3rd year) (experimental arm). Imatinib (Glivec), or Nilotinib (Tasigna), or Dasatinib (Sprycel) will be given intermittently at the same daily dose that was given daily at the time of the enrollment . Chronic phase Ph+ CML patients in stable major molecular response (MR3.0 or MR4.0) after ≥2 years of standard treatment with IM, NIL, or DAS will be randomized 1:1 to receive "fixed" INTERIM or "progressive" INTERIM. Randomization will be stratified by type of TKI (IM, NIL, or DAS,) and by depth of molecular response (MR3.0or MR4.0). The study is aimed to evaluate if a progressive increase of intermittent treatment discontinuation until 3 months is able to improve QoL outcomes with respect to "fixed" intermittent administration of TKIs (control arm) and to maintain MR3.0 / MR4.0 molecular response. Patients' self reported EORTC QLQ-C30 outcome measure will be assessed throughout the three years follow up period. The QoL results in this trial will be presented in accordance with high methodological quality criteria for documenting patient-reported outcomes (PRO) data in RCTs, including the CONSORT PRO recommendations. Furthermore, the study could give additional clinical and biological information to optimize TKIs therapy in elderly.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a confirmed diagnosis of Ph+ CML in CP
2. Age ≥ 60 years old
3. Stable MR3.0/ MR4.0 after at least 2 years of treatment with standard (daily administration) IM, NIL, or DAS therapy; the stability of molecular response will be documented by at least 3 consecutive molecular analyses over the last 12 months.
4. Having completed the QoL baseline evaluation (i.e., before randomization)
5. Written informed consent prior to any study procedures

Exclusion Criteria:

1. Patients with Ph+ CML in accelerated/blastic phase (AP/BP), or in late CP previously treated (i.e. IFNalpha+/- low dose Ara-C, Hydroxurea, allogeneic stem cell transplantation, etc)
2. Age < 60 years old
3. Less than 2 years of treatment with standard (continuous administration) IM, NIL or DAS therapy

3. Absence of stable MR3.0/MR4.0 as documented by at least 3 consecutive molecular analyses over the last 12 months 4. No written informed consent prior to any study procedures. 5. Having any kind of psychiatric disorder or major cognitive dysfunction hampering a QoL evaluation (as judged by the physician).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2015-06-10 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
Change in quality of Life | Baseline (T0), and then at 3 (T1), 6 (T2), 9 (T3), 12 (T4), 18 (T5), 24 (T6), 30 (T7), and 36 (T8) months

CONTACTS AND LOCATIONS:
Overall Officials: Domenico Russo, Professor, Principal Investigator — Chair of Hematology, BMT Unit
Locations (1):
- Policlinico Universitario di Milano, Milan, Italy